### **Informed Consent Form**

Title of Project: A Message Framing Intervention for Increasing Parental Acceptance of Human Papillomavirus Vaccination
NCT #: NCT03856437
02/10/2021

## Participant Consent Form

# **Project Title**

The HPV Vaccine Study

# Purpose of the Study

This research is being conducted by Dr. Xiaoli Nan and her research team at the University of Maryland, College Park. We are inviting you to participate in this research project because you 1) are at least 18 years old; 2) self-identify as African American; 3) are a custodial parent or caretaker of at least one child under the age of 18 who has not initiated or completed the HPV vaccine series. The purpose of this research project is to understand African American parents' responses toward HPV vaccination messages.

#### **Procedures**

The procedures involve completing a 20-minute computer-assisted survey. First you will answer questions related to your beliefs about HPV and the HPV vaccine, as well as other background information. Then you will be presented with a HPV vaccination message. After the message exposure, you will answer questions related to your attitudes toward HPV vaccination, intentions to vaccinate their children, as well as other message response measures. Sample questions include "how likely would you be to get your child vaccinated against HPV?" "what's your overall attitude toward HPV vaccination?"

## **Potential Risks and Discomforts**

There are no known risks associated with this research. Some participants may feel slightly uncomfortable answering some questions. All participants have the option of not responding to questions they do not wish to answer by exiting the study.

#### **Potential Benefits**

There are no direct benefits to you. However, we hope that, in the future, other people might benefit from this study through health communicators' improved understanding of how health messages are being perceived by the target audience, which, in turn, will lead to better health interventions.

## **Confidentiality**

Any potential loss of confidentiality will be minimized by storing data in a password protected computer in a locked office. For an online survey, we will immediately delete any identifying information like IP address after the data have been collected. Only approved researchers will have access to the data you provide. If we write a report or article about this research project, your identity will be protected to the maximum extent possible. Your information may be shared with representatives of the University of Maryland, College Park or governmental authorities if you or someone else is in danger or if we are required to do so by law.

## **Informed Consent Form**

Title of Project: A Message Framing Intervention for Increasing Parental Acceptance of Human Papillomavirus Vaccination
NCT #: NCT03856437
02/10/2021

### **Right to Withdraw and Questions**

Your participation in this research is completely voluntary. You may choose not to take part at all. If you decide to participate in this research, you may stop participating at any time. If you decide not to participate in this study or if you stop participating at any time, you will not be penalized or lose any benefits to which you otherwise qualify. If you decide to stop taking part in the study, if you have questions, concerns, or complaints, or if you need to report an injury related to the research, please contact the investigator: Dr. Xiaoli Nan, Department of Communication, University of Maryland, 2102 Skinner Building, 4300 Chapel Ln., College Park, MD 20742; email: nan@umd.edu; tel: 301-405-0640.

#### **Participants Rights**

If you have questions about your rights as a research participant or wish to report a research related injury, please contact:

University of Maryland College Park Institutional Review Board Office 1204 Marie Mount Hall College Park, Maryland, 20742 E-mail: irb@umd.edu

Telephone: 301-405-0678

This research has been reviewed according to the University of Maryland, College Park IRB procedures for research involving human subjects.

### **Statement of Consent**

Your online consent by clicking the radio button below indicates that you are at least 18 years of age; you have read this consent form or have it read to you; your questions have been answered to your satisfaction and you voluntarily agree to participate in this research study.

If you agree to participate, please choose the radio button "I agree to participate in this study" below.